CLINICAL TRIAL: NCT07219394
Title: Hybrid Effectiveness-Implementation Trial to Evaluate a Scalable, Peer-Delivered Intervention for Depression Among People With Substance Use Disorder in a Certified Community Behavioral Health Clinic
Brief Title: Peer-Delivered Behavioral Activation in a CCBHC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Julia Felton, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BARCT: 25-02-7552
Record Dates: First submitted 2025-07-21; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder; Substance Use Disorders
MeSH Terms: conditions — Depressive Disorder, Major; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Activation (Experimental): Peer Activate is an adapted behavioral activation (BA) intervention, developed for delivery by peer recovery specialists to reduce rates of depressive symptoms and substance use. BA focuses on increasing positive reinforcement through engaging in adaptive, valued behaviors. BA has been found to be effective in improving substance use outcomes and decreasing depressive symptoms among low-income individuals with SUD. Peer Activate includes 6 weekly sessions with up to 6 additional booster sessions.
  Interventions: Behavioral: Peer Activate
- Enhanced Treatment as Usual (Active Comparator): Enhanced treatment as usual (ETAU) involves peer-delivered non-directive support, including facilitated linkages to care and non evidence-based intervention approaches typically used by peer recovery specialists.
  Interventions: Behavioral: Peer-delivered non-specific services

INTERVENTIONS:
Behavioral: Peer Activate — Peer Activate is an adapted behavioral activation (BA) intervention, developed for delivery by peer recovery specialists to reduce rates of depressive symptoms and substance use. BA focuses on increasing positive reinforcement through engaging in adaptive, valued behaviors. BA has been found to be effective in improving substance use outcomes and decreasing depressive symptoms among low-income individuals with SUD. Peer Activate includes 6 weekly sessions with up to 6 additional booster sessions.
  Arms: Behavioral Activation
Behavioral: Peer-delivered non-specific services — Peers will deliver non-specific peer services, including linkage to care, general support, and facilitated referrals to external providers as needed.
  Arms: Enhanced Treatment as Usual

SUMMARY:
Low-income individuals have limited access to evidence-based interventions for mental health. Peer recovery specialists, individuals in recovery from mental health and/or substance use problems, have the potential to increase access to evidence-based interventions for individuals from low-resource communities, particularly when trained and supervised in models that are acceptable and feasible in these communities. This study will examine the effectiveness and implementation potential of a peer-delivered evidence-based intervention (Behavioral Activation) among individuals receiving services from a community-based treatment setting providing integrated physical and behavioral healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Report clinically-significant symptoms of depression, as indexed by a score of 8+ on the PHQ-9.

Exclusion Criteria:

* Active, under treated psychotic symptoms or mania that would interfere with participation in study procedures
* Inability to provide informed consent and/or complete procedures in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale | Baseline, post-intervention (approximately 3 months after baseline), 6- and 12-month follow-up
  The Hamilton Depression Rating Scale (HAM-D) is a structured interview regarding patients' symptoms of depression and functional impairment. The HAM-D will be administered by research assistants under the supervision of the MPI (Felton) at baseline, post-intervention, 6- and 12-month follow-up. The measure is widely used in depression and substance use treatment studies and has excellent psychometric properties. Nine items are scored 0-4 and 8 items are scored 0-2, with higher scores reflecting greater levels of depressive symptoms. A total score will be calculated by summing each other items. Summed total scores can range from 0-52, with higher values reflecting greater depression.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 | Baseline, post-intervention (approximately 3 months after baseline), 6- and 12-month follow-up
  The Patient Health Questionnaire-9 (PHQ-9) is a self-report measure of depressive symptoms. Participants will complete the PHQ-9 at baseline, post-intervention, 6- and 12-month follow-up. The measure is valid and reliable in low-resource community settings. The measure includes nine items which are scored from 0-3, with 3 reflecting more severe levels of each depressive symptom. A total score is created by summing items with a possible range from 0-27 (with higher scores reflecting greater depressive symptoms).
Change in Short Inventory of Problems | Baseline, post-intervention (approximately 3 months after baseline), 6- and 12-month follow-up
  The Short Inventory of Problems is a self-report measure of problems related to substance use. Participants will complete the SIP at baseline, post-intervention, 6- and 12-month follow-up. The measure is valid and reliable and has been used by the investigator team in numerous studies among low-income populations. The measure includes 17 items, each ranked from 0-3 with higher scores reflecting greater problems related to alcohol and substance use. A total score is created by summing each item and can range from 0-51 with higher values reflecting more substance-related problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Recovery Project, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No